CLINICAL TRIAL: NCT01621035
Title: Objective Assessment of Physical Activity in Older Adults
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML7732
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Functionality; Strength; Validity During Daily Activities; Physical Activity; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- elderly (> 70 y)

SUMMARY:
The purpose of the present study is to evaluate the validity of 2 objective measures of physical activity among older adults. In addition, the investigators will examine the influence of functionality, walking aids, walking speed and step length on the accuracy.

ELIGIBILITY:
Inclusion Criteria:

* > 70 years

Exclusion Criteria:

* recent cardiovascular event
* vestibular disorder or fracture (4 months)
* severe dementia
* oxygen supplementation during daily activities
* not able to perform daily activities

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults (> 70 years)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Leuven, Belgium